CLINICAL TRIAL: NCT00562731
Title: A Phase III, Open-Label Follow-on Study for Long-Term Safety and Efficacy of Testosterone Cream, in Testosterone Deficinet Men Completing Study ARD-0403-004
Brief Title: Open-Label Study of ARD-0403 in Testosterone Deficient Men
Acronym: ARD-0403-010
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company strategic decision
Sponsor: Ardana Bioscience Ltd (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARD-0403-010
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism

INTERVENTIONS:
Drug: ARD-0403 — Daily transdermal ARD-0403

SUMMARY:
Male hypogonadism, a disorder associated with testosterone deficiency, is frequently seen in clinical practice and has significant effects on patient well-being. The purpose of this study is to investigate the efficacy and safety of ARD-0403 as a testosterone replacement therapy in testosterone deficient men.

ELIGIBILITY:
Inclusion Criteria:

* Testosterone deficiency
* Completed study ARD-0403-004

Exclusion Criteria:

* Previous treatment with testosterone replacement therapy within 4 weeks
* Moderate-severe benign prostatic hypertrophy or prostatic cancer
* Haematocrit >50%

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-10; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy | Study Duration

SECONDARY OUTCOMES:
Safety and Tolerability | Study Duration

CONTACTS AND LOCATIONS:
Overall Officials: R Swerdloff, Principal Investigator — University of California, Los Angeles
Locations (12):
- United States (12):
  - Medical Affiliated Research Center, Inc, Huntsville, Alabama
  - Stanford University, Stanford, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - dgd Research, San Antonio, Texas
  - VA Puget Sound Health Care System, Seattle, Washington